CLINICAL TRIAL: NCT04788654
Title: The Comparison of Multimodal Analgesic Protocols for Laparoscopic Cholecystectomy: Pharmacologic Interventions and Combination of Pharmacologic and Operative Interventions
Brief Title: Multimodal Analgesia for Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Do-Hyeong Kim, Associate professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3-2020-0494
Record Dates: First submitted 2021-02-16; First posted 2021-03-09 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib; Acetaminophen; Dexamethasone; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacological group (Active Comparator): Pharmacological analgesia will be performed
  Interventions: Drug: Celebrex, acetaminophen, and dexamethasone
- Pharmacologican and surgical group (Experimental): Pharmacological and surgical analgesia will be performed.
  Interventions: Drug: Celebrex, acetaminophen, and dexamethasone; Procedure: Saline irrigation, aspiration of pneumoperitoneum, and low pressure penumoperitoneum

INTERVENTIONS:
Drug: Celebrex, acetaminophen, and dexamethasone — Pharmacological intervention will be performed. Celebrex 200mg, acetaminophen 1g, and dexamethasone 7 mg will be infused perioperatively.
  Other Names: Pharmacological
Procedure: Saline irrigation, aspiration of pneumoperitoneum, and low pressure penumoperitoneum — Surgical intervention will be performed. Saline irrigation, aspiration of pneumoperitoneum, and low pressure pneumoperitoneum will be performed.
  Other Names: Surgical
  Arms: Pharmacologican and surgical group

SUMMARY:
It is important to decrease the postoperative pain in patients undergoing laparoscopic cholecystectomy. We will compare the pharmacologic analgesia with the parmacologic and surgical analgesia in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3, and scheduled for elective laparoscopic cholecystectomy

Exclusion Criteria:

1. Recent gastric ulcer disease
2. Hepatic or renal insufficiency
3. Opioid dependency
4. Coagulopathy
5. Pre-existing neurologic or anatomic deficits in the lower extremities
6. Severe psychiatric illness
7. pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Area under curve of postoperative pain for 24 hour | At postoperative 24 hour
  Area under curve will be measured using Postoperative pain score at postoperative 24 hour using visual anlogue scale (0: no pain, 10: most imaginable pain).

SECONDARY OUTCOMES:
Postoperative pain score, | At postoperative 0, 2, 6, and 24 hour
  Postoperative pain score: postoperative pain score will be measured at postoperative 0, 2, 6, and 24 hour using visual anlogue scale (0: no pain, 10: most imaginable pain).
Analgesic requirements, | At postoperative 24 hour
  Analgesic requirements will be measured at postoperative 24 hour. Total dose of tramadol, ketorolac, and pethidine will be assessed at postoperative 24 hour.
Sleep quality | At postoperative 24 hour
  Sleep quality will be measured using sleep quality questionnare at postoperative 24 hour.
  using sleep quality questionnare.

CONTACTS AND LOCATIONS:
Locations (1):
- Do-Hyeong Kim, Seoul, South Korea